CLINICAL TRIAL: NCT03144843
Title: A Phase II Multicenter, Randomized, Double-blind Study of Apatinib Combined With Paclitaxol Versus Placebo With Paclitaxol as Second Line Therapy for Advanced Gastric / Esophagogastric Junction Adenocarcinoma With Peritoneal Metastasis.
Brief Title: Apatinib Combined With Paclitaxol as Second Line Therapy for Advanced Gastric Cancer.
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Collaborators: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Fenghua Wang, Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Apatinib_GC
Record Dates: First submitted 2017-05-05; First posted 2017-05-09 (Actual); Last update posted 2017-05-09 (Actual); Status verified 2017-05

CONDITIONS: Gastric Cancer
Keywords: Gastric cancer; Peritoneal metastasis; Paclitaxol; Apatinib; Second-line chemotherapy
MeSH Terms: conditions — Stomach Neoplasms | interventions — apatinib

STUDY DESIGN:
Intervention Model Description: Multicenters ramdomized double-blind phase II study.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Apatinib: 500mg, po, qd, every 4 weeks Paclitaxol: 80mg/m2, d1, d8, d15, every 4 weeks
  Interventions: Drug: Apatinib
- Placebo group (Placebo Comparator): Placebo: 500mg, po, qd, every 4 weeks Paclitaxol: 80mg/m2, d1, d8, d15, every 4 weeks
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Apatinib — Apatinib 500mg, po, qd, every 4 weeks Paclitaxol: 80mg/m2, d1, d8, d15, every 4 weeks
  Other Names: Paclitaxol
  Arms: Experimental group
Drug: Placebos — Placebo: 500mg, po, qd, every 4 weeks Paclitaxol: 80mg/m2, d1, d8, d15, every 4 weeks
  Other Names: Paclitaxol
  Arms: Placebo group

SUMMARY:
This multicenter, randomized, double-blind study will evaluate the efficacy and safety of apatinib combined with paclitaxol versus placebo combined with paclitaxol in advanced gastric cancer or gastroesophageal junction carcinoma patients with peritoneal metastasis.

Patients will be randomized to one treatment arm: Arm A: apatinib 500mg qd, Paclitaxol 80mg/m2, d1, d8, d15,every 4 weeks ; Arm B: placebo 500mg qd, Paclitaxol 80mg/m2, d1, d8, d15,every 4 weeks ; Tumor assessment will be done every 8 weeks according to RECIST 1.1. The primary endpoint is progression free survival (PFS).

DETAILED DESCRIPTION:
Gastric cancer is the second most common cause of cancer-related deaths worldwide, and most patients are diagnozed at advanced stage in China. Peritoneal metastasis is the most common metastatic site. For gastric cancer patients with peritoneal metastasis, chemotherapy can bring survival benefit versus best sportive care. Paclitaxol is the standard second line chemotherapy for advanced gastric cancer patients.

Apatinib mesylate is a small-molecule vascular endothelial growth factor receptor-2 (VEGFR-2) tyrosine kinase inhibitor (TKI). It has been approved as third-line treatment for patients with advanced gastric adenocarcinoma in China.

This multicenter, randomized, double-blind study will evaluate the efficacy and safety of apatinib combined with paclitaxol versus placebo combined with paclitaxol in advanced gastric cancer or gastroesophageal junction carcinoma patients with peritoneal metastasis.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients, aged between 18 and 75 years old;
2. Histologically confirmed advanced or metastatic adenocarcinoma of gastric cancer(AGC) , including adenocarcinoma of the gastroesophageal junction ;
3. At least one measurable and evaluable disease based on response evaluation criteria in solid tumors (RECIST v1.1); and confirmed as peritoneal metastasis by CT scan or laparoscope
4. Patients must have received one prior chemotherapy regimen for AGC;First-line therapy must have included a combination of at least a platinum-based treatment given concurrently, and must have experienced disease progression during or after first-line therapy for their disease;
5. Eastern Cooperative Oncology Group(ECOG) performance status of 0 or 1;
6. Life expectancy of more than 3 months;
7. Duration from the last therapy is more than 6 weeks for nitroso or mitomycin, More than 4 weeks for other cytotoxic agents, operation or radiotherapy;
8. Adequate hepatic, renal, heart, and hematologic functions ( hemoglobin≥ 90g/L, platelets ≥ 80 × 10*9/L, neutrophil ≥1.5 × 10*9/L, serum creatinine≤ 1.5mg/dl, total bilirubin ≤1.5 ×ULN, and serum transaminase≤2.5×ULN)

Exclusion Criteria:

1. Pregnant or lactating women;
2. History of other malignancies except cured basal cell carcinoma of skin and carcinoma insitu of uterine cervix;
3. Prior chemotherapy regimen have included taxane (docetaxel or paclitaxel); 4. Uncontrolled hypertension;

5. Intercurrence with one of the following: coronary artery disease, arrhythmia and heart failure; 6. Urine protein>grade 1; 7. Any factors that influence the usage of oral administration; 8. Patients with a clear tendency of gastrointestinal bleeding; 9. Abnormal coagulation function(INR≥1.5, APTT≥1.5 ULN); 10. Abuse of alcohol or drugs; 11. Less than 4 weeks from the last clinical trial; 12. Prior treatment with antivascular endothelial growth factor or the other anti angiogenesis therapy; 13. Evidence of central nervous system(CNS) metastasis; 14. Disability of serious uncontrolled intercurrence infection.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2017-01-13 (Actual); Primary Completion 2020-01-31 (Estimated); Study Completion 2020-01-31 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | Approximately 1 year
  The time from randomize to progression or death

SECONDARY OUTCOMES:
Overall survival (OS) | Approximately 3 years
  The time from randomize to death
Objective response rate (ORR) | Approximately 1 year
  The rate of complete response and partial response according to RECIST guidelines
Disease control rate(DCR) | Approximately 1 year
  The rate of complete response , partial response and stable disease according to RECIST guidelines
Safety (incidence of adverse events) [ | Approximately 1 year
  Incidence of adverse events

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Foshan people's Hospital, Foshan, Guangdong
  - Cancer center of Sun Yat-sen University, Guangzhou, Guangdong

IPD SHARING:
Plan to Share IPD: No